CLINICAL TRIAL: NCT06062264
Title: Improving Influenza Vaccination Delivery Across a Health System by the Electronic Health Records Patient Portal RCT 6
Brief Title: Patient Portal Flu Vaccine Reminders (RCT 6)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Executive Vice Chair, Vice Chair for Research, UCLA David Geffen School of Medicine, Department of Pediatrics, University of California, Los Angeles, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-001889-00018; R01AI135029 (NIH)
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Influenza; Respiratory Tract Infections
Keywords: Reminder Recall (R/R); Influenza Vaccine; Electronic Health Record; Vaccine; Video Messages; Trusted Messenger
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Pragmatic comparative effectiveness trial with a standard-of-care control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Portal-Based PCP Video Reminder Message (Active Comparator): Participants in their arm will receive up to 3 portal-based messages with a video recorded message from their own primary care physician encouraging them to receive the influenza vaccine.
  Interventions: Behavioral: Portal-based Video Message
- Portal-Based PCP Infographic Reminder Message (Active Comparator): Participants in their arm will receive up to 3 portal-based messages with an infographic message with an image of their own primary care physician encouraging them to receive the influenza vaccine.
  Interventions: Behavioral: Portal-based Infographic Message
- Standard Health System Portal Messages (No Intervention): Participants in this arm will only receive standard-of-care health system portal messages, and will not receive study-based messages.

INTERVENTIONS:
Behavioral: Portal-based Video Message — Video recorded by physician encouraging patients to receive influenza vaccine. Sent via the patient portal.
  Arms: Portal-Based PCP Video Reminder Message
Behavioral: Portal-based Infographic Message — Infographic with information about the influenza vaccine and an image of the physician. Sent via the patient portal.
  Arms: Portal-Based PCP Infographic Reminder Message

SUMMARY:
This trial is taking place in Los Angeles, CA at 21 clinics within the UCLA Health System.

The study design is a 3 arm randomized trial. Patients will be randomized into 1) receiving portal based reminder messages with a video from their PCP encouraging them to receive the influenza vaccine, 2) portal-based reminder messages with an infographic with the image of their PCP encouraging them to receive the influenza vaccine, or 3) the control group. Patients randomized to the intervention arms will receive reminders if they are due for influenza vaccine.

Despite the Advisory Committee on Immunization Practices (ACIP) recommendation in 2010 that all people above 6 months of age should receive an annual flu vaccine, vaccination rates remain low: at 6m-4.9 yrs. (70%), 5-17.9 yrs. (56%), 18-64.9 yrs. (38%), and >65 yrs. (63%). The investigators will assess the effectiveness of MyChart R/R video messages and infographic messages as compared to the standard of care control (Health system messages).

DETAILED DESCRIPTION:
Sub-optimal vaccination rates are a significant problem in the U.S., despite their effectiveness in preventing morbidity and mortality from vaccine-preventable illness. For influenza specifically, annual epidemics of influenza cause substantial morbidity in the U.S. with up to 40,00-80,000 deaths/year and many hospitalizations, emergency and outpatient visits, and significant costs.

Reminder/recall (R/R), sent by phone, mail or other modality, can improve child and adult influenza vaccination rates. However, the majority of pediatric or adult primary care practices do not conduct R/R. Barriers are lack of finances, personnel, and algorithms to identify eligible patients.

A technological breakthrough that might overcome these barriers involves patient portals-- secure, web-based communication systems, embedded within electronic health records (EHRs), for patients and providers to communicate with each other via email and the internet. Portals are used by about half of Americans and half of UCLA patients. Another is text messaging at the health system level.

This randomized controlled trial will assess the effectiveness of reminders messages sent to portal users, encouraging influenza vaccination, on increasing influenza vaccination rates within a health system. Patients will be randomized into three groups: 1) one-third of patients will receive reminder messages with a video from their PCP encouraging them to receive the influenza vaccine, 2) one-third will receive reminders with an infographic with information about the influenza vaccine with an image of their PCP, and 3) one-third will receive standard health system messages (standard of care).

Portal-based video messages: Clinicians have been shown to be trusted by their patients, so by sending patients videos that have been recorded by their own primary care physician, we are testing the concept of 'trusted messengers' to improve influenza vaccine uptake.

Portal-based infographic messages: This study arm is also testing the concept of 'trusted messenger' since all infographic messages will also have an image of patients' own primary care physician at the top.

Interventions that apply Behavioral Economics principles in vaccine promotion messaging can increase vaccine receipt. In the physician videos and infographics we will also include language utilizing the concepts endorsing social norms, social good, positive framing, urgency, and planning.

For the primary analysis, the primary outcome will be the patient's end of flu season vaccination status. Intervention effects will be assessed using mixed effects log-binomial models.

The portal-based reminder messages will be sent in October of 2023. Repeat messages will also be sent in late October, and late November to patients who do not receive their influenza vaccines.

ELIGIBILITY:
Inclusion Criteria:

- Active Portal Users A patient within the UCLA Health System identified as a primary care patient per an internal algorithm

Exclusion Criteria:

- A patient within the UCLA Health System not identified as a primary care patient per an internal algorithm

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22233 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szilagyi, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Szilagyi PG, Clark EJ, Duru OK, Casillas A, Ong MK, Vangala S, Tseng CH, Albertin C, Humiston SG, Ross MK, Evans S, Kumar A, Chakarian I, Sloyan M, Fox CR, Rand CM, Lerner C. Video and Infographic Messages From Primary Care Physicians and Influenza Vaccination Rates: A Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2526514. doi: 10.1001/jamanetworkopen.2025.26514. PMID 40802184

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Portal-Based PCP Video Reminder Message | Portal-Based PCP Infographic Reminder Message | Standard Health System Portal Messages
Started | 7410 | 7406 | 7417
Completed | 7410 | 7406 | 7417
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Portal-Based PCP Video Reminder Message | Portal-Based PCP Infographic Reminder Message | Standard Health System Portal Messages | Total
Number analyzed (Participants) | 7410 | 7406 | 7417 | 22233
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1058 | 1085 | 1057 | 3200
  Between 18 and 65 years | 4908 | 4915 | 4881 | 14704
  >=65 years | 1444 | 1406 | 1479 | 4329
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4647 | 4658 | 4668 | 13973
  Male | 2763 | 2748 | 2749 | 8260
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 776 | 795 | 843 | 2414
  Black | 326 | 352 | 338 | 1016
  White | 3797 | 3618 | 3635 | 11050
  Other (Unknown or Multiple) | 2511 | 2641 | 2601 | 7753
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 1020 | 1008 | 1044 | 3072
  Non-Hispanic or Unknown | 6390 | 6398 | 6373 | 19161
Primary Insurer [Count of Participants; unit: Participants]
  Private | 6307 | 6302 | 6269 | 18878
  Public | 996 | 996 | 1035 | 3027
  Other/Unknown/Multiple | 107 | 108 | 113 | 328
Influenza Vaccine History [Count of Participants; unit: Participants]
  None | 1949 | 1974 | 1964 | 5887
  Prior Vaccination | 5461 | 5432 | 5453 | 16346

OUTCOME MEASURES:

1. Primary Outcome: Receipt of the Annual Influenza Vaccine Among Index Patients
Description: Percent of patients with annual influenza vaccination (between 10/4/23 - 4/1/24) among adult patients. Outcomes will be assessed via vaccine data extraction from the electronic health record and external claims and pharmacy data.
  The index patients must also be an active UCLA Health MyChart user (>= 1 login over the last 12 months from 8/1/23, excluding activity on the user's initial profile activation date). Individuals not affiliated with any primary care practice will be excluded from the primary analysis.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Portal-Based PCP Video Reminder Message | Portal-Based PCP Infographic Reminder Message | Standard Health System Portal Messages
Number analyzed (Participants) | 7410 | 7406 | 7417
Participants | 3557 | 3518 | 3479
Statistical Analysis 1: Comparison: Portal-Based PCP Video Reminder Message vs Standard Health System Portal Messages; Comparing the risk of receiving an influenza vaccination; Test type: Superiority; Adjusted Risk Ratio = 1.03, 95% CI 2-sided [1.00 to 1.06]; Adjusted risk ratio. These results compare arms which received portal-based PCP video reminder messages to the arm receiving standard health system portal messages (control)
Statistical Analysis 2: Comparison: Portal-Based PCP Infographic Reminder Message vs Standard Health System Portal Messages; Comparing the risk of receiving an influenza vaccination; Test type: Superiority; Adjusted Risk Ratio = 1.02, 95% CI 2-sided [0.99 to 1.06] — Adjusted risk ratio. These results compare arms which received portal-based PCP video reminder messages to the arm receiving standard health system portal messages (control)

2. Secondary Outcome: Receipt of the Annual Influenza Vaccine Among Pediatric Index Patients
Description: Percent of patients with annual influenza vaccination (between 10/4/23 - 4/1/24) among pediatric index patients. Outcomes will be assessed via vaccine data extraction from the electronic health record and external claims and pharmacy data.
  The index patients must also be an active UCLA Health MyChart user (>= 1 login over the last 12 months from 8/1/23, excluding activity on the user's initial profile activation date). Individuals not affiliated with any primary care practice will be excluded from the primary analysis.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Portal-Based PCP Video Reminder Message | Portal-Based PCP Infographic Reminder Message | Standard Health System Portal Messages
Number analyzed (Participants) | 1058 | 1085 | 1057
Participants | 618 | 598 | 576

ADVERSE EVENTS:
Time Frame: We did not collect information regarding adverse events or deaths.
Description: We did not collect adverse event or death information. We monitored whether reminder recall through the portal and text was effective at increased influenza vaccination rates. Because influenza vaccination is recommended by the Advisory Committee on Immunization Practices and is part of the U.S. recommended vaccine schedule, we did not collect adverse event data.
Arm/Group | Portal-Based PCP Video Reminder Message | Portal-Based PCP Infographic Reminder Message | Standard Health System Portal Messages
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT06062264/Prot_SAP_000.pdf